CLINICAL TRIAL: NCT06206317
Title: Comparison of Motor and Sensory Functions of the Hand in Children With Type 1 Diabetes Mellitus and Their Healthy Peers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erdal AYDIN (Other)
Responsible Party: Sponsor-Investigator, Erdal AYDIN, Principal Investigator, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Other Study IDs: erdalaydin.T1DM
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus (T1DM); Hand Grip Strength; Fine Grip Strength; Semmes-Weinstein Monofilaments; Sensation of the hand; hand functions; Pediatric Endocrinology Clinic; Vibration Sensation; Static Two-Point Discrimination; Functional Skills Test; Jebsen Taylor Hand Function Test (JTEFT)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Comprising children diagnosed with Type 1 Diabetes Mellitus (T1DM). This group constitutes the focal point of the study, assessing the motor and sensory functions of the hand. These children undergo various tests and measurements aimed at evaluating the motor skills, sensory perception, and functionality of the hand. The study solely involves evaluation and will not include any treatment or intervention.
- Control Group: Consisting of children without any health issues. This group comprises healthy individuals and serves as a comparative reference against the study group. Similar tests and measurements are applied to assess the motor and sensory functions of the hand in healthy individuals for comparison with the study group. The study solely involves evaluation and will not include any treatment or intervention.

SUMMARY:
Type 1 Diabetes Mellitus (T1DM) is a condition where the body cannot produce a hormone called insulin. Although it is commonly seen in children and young people, it can occur at any age. The effects of T1DM on hand functions in children, particularly, have not been thoroughly researched yet. However, studies indicate that children diagnosed with diabetes may experience weakness in wrist muscles, reduced sensitivity in fingers, and impaired hand coordination. This study aimed to compare the motor and sensory functions of hands in children with T1DM against healthy children.

This study will compare children with T1DM to healthy children. Children will be divided into two groups: one group comprising children with T1DM, and the other including healthy children with no medical conditions. Children between the ages of 7-18 diagnosed with T1DM will participate in the study. The healthy control group will consist of children without any health issues within the same age range who visit the hospital for routine check-ups. In total, 140 children will be included in the study, with 70 children having diabetes and 70 healthy children.

Tests used in the study:

* The Jebsen Taylor Hand Function Test (JTEFT) is a standard test used to assess hand functions, consisting of 7 different sub-tests.
* The Functional Skill Test (FBT) is utilized to evaluate children's fine motor skills.
* Handgrip strength will be measured using the jamar hydraulic Hand Dynamometer.
* Fine grip strength is assessed using a device called Baseline®, measuring finger grip strength with different grips.
* Semmes-Weinstein monofilaments (SWM) are used to test light touch/pressure sensation. *Monofilaments are applied to specific points, determining the lightest pressure level the patient feels.
* A discriminator is used for static two-point discrimination measurement, testing whether the patient can feel two separate points.
* Vibration sensation is measured by touching at a specific frequency.
* For Hot-Cold Assessment, tubes with different temperature water are used, and the person is asked to identify which tube feels hot or cold.

DETAILED DESCRIPTION:
Type 1 Diabetes Mellitus (T1DM) is a metabolic disorder characterized by complete insulin deficiency, typically resulting from the destruction of beta cells, and identified by elevated blood sugar levels. T1DM is commonly observed in children and adolescents but can occur at any age. Microvascular complications such as visual impairment, kidney disease, neuropathy, and diabetic foot ulcers can arise in individuals with T1DM. Various musculoskeletal disorders like Dupuytren's syndrome, osteoporosis, osteopenia, adhesive capsulitis, carpal tunnel syndrome, and limited joint mobility syndrome can also be observed in individuals with T1DM. Limited joint mobility syndrome has been reported in 38-58% of type 1 diabetic patients, showing increased stiffness in the hand. The increased stiffness in the hand leads to fixed flexion contracture in the hand joints, disrupting fine motor skills and grip strength. The Semmes-Weinstein monofilament examination can predict foot ulceration and amputation risk in diabetic patients and aid in detecting diabetic peripheral neuropathy. Vibration testing, along with the Semmes-Weinstein monofilament examination, can detect diabetic peripheral neuropathy. A study by Hirschfeld et al. indicated that vibration testing exhibits high specificity for detecting diabetic peripheral neuropathy in children and adolescents. In a study conducted by Ising et al. in 2018, altered vibrotactile sensation indicative of diabetic peripheral neuropathy was found in 1/5 of adolescents and children. Reduced joint mobility in the hand, along with sensory loss, can also lead to decreased grip strength. A condition associated with insulin resistance and glucose metabolism in adolescents has been linked to grip ability. According to American Diabetes Association (ADA), individuals diagnosed with T1DM should be screened for diabetic peripheral neuropathy annually, starting within five years of the T1DM diagnosis. These screenings should assess thermal discrimination, vibratory sensation using a 128-hertz (Hz) tuning fork, and light touch sensation using a 10g monofilament test to determine ulceration and amputation risk.

Objective of our study: To compare the motor and sensory functions of the hand in children diagnosed with Type 1 Diabetes Mellitus with those of healthy peers.

Materials and Methods:

This study will be conducted at the Pediatric Endocrinology Clinic of Health Practice and Research Hospital. Participants will be divided into two groups: a study group consisting of individuals diagnosed with T1DM and a control group without any health issues. The study group will include children aged 7-18 years who have been diagnosed with T1DM and are seeking care at the pediatric endocrinology clinic. The control group will comprise children aged 7-18 years without any health problems, attending the hospital for routine check-ups or accompanying family members. The study will include 70 children diagnosed with T1DM and 70 healthy children, totaling 140 participants. The control group will be age-matched with the study group. Demographic information will be collected after obtaining written and verbal consent from the participants. Motor and sensory assessments of the hand will be conducted and compared.

Tests used for hand sensory, motor, and functional assessment:

*Jebsen Taylor Hand Function Test (JTEFT) is a standardized test developed by Jebsen et al. in 1969, comprising seven sub-tests to evaluate hand functions objectively. The test demonstrates high reliability and validity, with reference values prepared for different age groups and genders.

The sub-tests include:

1. Writing a sentence (24 words) ("The Weather Will Be Cloudy With Rain")
2. Flipping 5 cards: (3x5 inches in size)
3. Small object retrieval and placing them into a tin box (2 paper clips, 2 coins, and 2 soda caps)
4. Using a dessert spoon to pick up 5 dried kidney beans (nutrition simulation)
5. Stacking backgammon stones (using a wooden backgammon piece)
6. Throwing 5 lightweight tin cans across a distance
7. Throwing 5 heavy tin cans (450g) across a distance The test is time-limited, with a time limit given for each sub-test. The time taken by the child to complete each sub-test is recorded in seconds. A shorter completion time indicates better performance. To ensure standardization, a scaled board among the test materials and a stopwatch for timing the activities are used. The chair and table used during the test should be of appropriate size for the child. Before administering the test, the child is instructed and shown how to perform the tasks. Explaining that the test is time-limited is necessary for the child's motivation. The child starts with a "begin" command, and when the child finishes the activity, the stopwatch is stopped. The time taken to complete each activity for both the dominant and non-dominant hand is recorded in seconds for scoring.

   * Functional Dexterity Test (FDT) provides information about fine motor skills in children. The examiner places a pegboard (a square board with 16 holes measuring 20.6 cm in one side) on the edge of a table where the child is seated. The researcher instructs the child to flip each peg (a wooden piece with one black and one red side) over. Starting from the farthest peg from the tested hand, the pegs are flipped in a zigzag pattern and then placed back onto the pegboard. The researcher uses a stopwatch to calculate the time taken to flip all pegs and records it in seconds. At the end of the study, two scores are obtained: the time taken to complete the test in seconds and the completion rate (rate = number of flipped pegs / seconds). Normative values for FDT are available for children aged 3 to 17.
   * Hand grip strength will be evaluated using a jamar Hydraulic Hand Dynamometer in the standardized test position established by the American Society of Hand Therapists. During measurement, the children will be positioned in a chair without back support, sitting upright. Measurements will be taken with the shoulder in adduction, the elbow at 90 degrees of flexion, the forearm in a neutral position, and the wrist in 0-30 degrees of extension and 0-15 degrees of ulnar deviation. Three measurements of muscle strength will be taken for both the right and left hands, and the average values will be recorded in kilograms. A 1-minute rest period will be given between each test.
   * Baseline® pinch gauge will be used for evaluating fine pinch grip strength. Measurements will be performed in the position defined by the American Society of Hand Therapists (the child sitting in a position without back support, with the shoulder in adduction, and the forearm and wrist in a neutral position). The child will be positioned so that the hips and knees are flexed at a 90° angle. Three measurements will be taken for each type of grip (lateral, palmar, and tip-to-tip). In the lateral grip, the midpoint of the thumb's distal phalanx is placed against the middle radial aspect of the index finger. In the palmar grip, the distal palmar surface of the thumb is placed against the distal palmar surfaces of the second and third fingers. In the tip-to-tip grip, the distal interphalangeal and proximal interphalangeal joints of the thumb and index finger are flexed, and their distal ends are brought together. The child will be instructed to exert the maximum force possible on the gauge for each grip position, followed by relaxation after each measurement. After three measurements in each position, a 15-second rest period will be given before testing the other hand. The results will be recorded in kilograms, and their average values will be calculated.
   * Semmes-Weinstein monofilaments (SWM) with values ranging from 1.65 to 6.65 will be used for evaluating light touch/pressure sensation. Three points will be tested in the areas innervated by the median and ulnar nerves: for the median nerve, the 1st fingertip, 2nd fingertip, and proximal phalanx of the 2nd finger; for the ulnar nerve, the 5th fingertip, proximal phalanx of the 5th finger, and proximal hypothenar area will be tested. The assessment starts with the lightest monofilament and progresses until the patient feels the monofilament. The tip of the monofilament is applied to the predetermined points for 1.5 seconds. Three assessments will be conducted, and at least 2 correct responses are required. If this condition cannot be met, the value of the monofilament used will be considered. The classification for SWM test results is as follows: 1.65-2.83 (green), normal sensation; 3.22-3.61 (blue), decreased light touch sensation; 3.84-4.31 (purple), decreased protective sensation; 4.56-6.65 (red), loss of protective sensation.
   * The static two-point discrimination test will be conducted using a discriminator. The two ends of the discriminator will be adjusted to a distance of 5 mm, and the child will be asked to indicate whether they feel one or two points. The discriminator will apply equal pressure to both ends simultaneously with a slight touch. Each test point will be touched three times with the discriminator. The distance where the child reports feeling one or cannot differentiate in two out of three tests will be recorded as the child's two-point discrimination score. The values obtained from the four test points will be added together and divided by four to calculate the average value.
   * Vibration sensation will be assessed using a 128 Hz tuning fork. During measurement, the child will be positioned in a chair without back support, sitting upright. The assessment will be performed with the shoulder in adduction, the elbow at 90 degrees of flexion, and the forearm in a neutral position while the child's eyes are closed. The assessment will be conducted on the second metacarpal head, the fifth metacarpal head, and the fingertip of the index finger. The duration of vibration sensation felt by the patient will be recorded using a stopwatch.
   * For the hot-cold assessment, two tubes containing hot and cold water, respectively, will be used. The temperature of the hot water will be set at 45 degrees Celsius, and the cold water at 25 degrees Celsius. To eliminate visual cues, the individual will be asked to look in a different direction. After contacting the dermatome area with the tubes, the person will be asked which tube contains hot or cold water. Scoring will be as follows: 1 point if the person correctly identifies the tubes and 0 points if they answer incorrectly.

Hypotheses of this study:

H0: There is no significant difference in the motor and sensory functions of the hand between children diagnosed with Type 1 Diabetes Mellitus and their healthy peers.

H1: There is a significant difference in the motor and sensory functions of the hand between children diagnosed with Type 1 Diabetes Mellitus and their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study.
* Being diagnosed with T1DM.
* The consent of the family for the study has been obtained and the consent document has been signed.
* Being between the ages of 7-18 years.
* To be co-operative during the evaluations.
* Not having orthopedic and neurological problems that prevent the evaluation.

Exclusion Criteria:

* Refusal to participate in the study.
* Parents have not signed a consent form.
* Not being between the ages of 7-18.
* Not being able to co-operate during the evaluations.
* Having orthopedic and neurological problems that prevent the evaluation.
* Having an additional disease (celiac, autoimmune disease, etc.)
* Not being able to comply with the researcher's commands during the evaluation

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will be conducted in the Pediatric Endocrinology Outpatient Clinic of Hatay Mustafa Kemal University, Health Practice and Research Hospital. The participants included in the study will be divided into 2 groups as the study group including those diagnosed with T1DM and the control group without any health problems. The study group will include children between the ages of 7-18 years who have been diagnosed with T1DM and who apply to the paediatric endocrinology outpatient clinic. In the control group; children between the ages of 7-18 years who agree to participate in the study, who do not have any health problems, who come to the hospital for control or who come to accompany their family members will be included.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-02-03 (Estimated); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength Measurement | 1 minute
  Jamar Hydraulic Hand Dynamometer is used to measure hand grip strength in a standardized test position defined by the American Society of Hand Therapists. Measurements are taken for both the right and left hands, and average values are recorded in kilograms.
Fine Grip Strength Assessment | 2 minute
  The "pinchmeter" is used to measure finger grip strength in lateral, palmar, and fingertip grasp positions. Three measurements are taken for each grip, and the results are recorded in kilograms.
Jebsen Taylor Hand Function Test (JTEFT) | 8 minute
  This test is utilized to evaluate hand functions. It includes activities such as writing a sentence, flipping cards, picking up and placing small objects in a container, picking up beans using a teaspoon, stacking checkers, tossing lightweight cans, and heavier cans. Each activity must be completed within a designated time frame. Results are derived from the time taken to complete the activities.
Functional Skills Test | 4 minute
  This test assesses fine motor skills. Using a pegboard, the child is instructed to turn over and place circular discs in sequence. The test measures completion time and speed.
Semmes-Weinstein Monofilament Examination | 4 minute
  This test evaluates light touch/pressure sensation using monofilaments of varying pressure values. Applied at three points in areas innervated by the median and ulnar nerves, the test results are classified within specific ranges to assess changes in sensory perception.
Vibration Test | 4 minute
  Vibratory sensation is measured using a 128 Hz diapason. The time taken by the patient to perceive the vibration applied to specific points is recorded using a stopwatch.
Hot-Cold Assessment | 2 minute
  Using two tubes containing hot and cold water, the patient's ability to distinguish between hot and cold is tested within the dermatomal area. Results are evaluated based on the accuracy of identifying the temperatures.
Static Two-Point Discrimination Test | 2 minute
  This test measures the ability to distinguish between two points applied simultaneously to the skin. A calibrated two-point discriminator is used to assess whether the individual can perceive whether it's one or two points being touched. The results are recorded based on the patient's ability to discern the two-point stimuli and are evaluated as the patient's two-point discrimination score. This test is an essential tool in assessing sensory capabilities in the hand.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Bezgin, Study Director — Mustafa Kemal University

IPD SHARING:
Plan to Share IPD: Undecided
No decision has been made as the work has not started yet.